CLINICAL TRIAL: NCT06054503
Title: A French Monocenter, Interventional Pilot Clinical Investigation to Evaluate the Technical Performance and Safety of a Prototype of Sensor to Measure Ventilator-derived Parameters in Intubated and Mechanically Ventilated Patients
Brief Title: Pilot Clinical Investigation to Evaluate a Prototype of Sensor Measuring Ventilator-derived Parameters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Archeon (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: H03
Record Dates: First submitted 2023-07-12; First posted 2023-09-26 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2023-09

CONDITIONS: Mechanically Ventilated Patients

STUDY DESIGN:
Intervention Model Description: The patient is his own control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- prototype of sensor (Experimental): The patient is his own control
  Interventions: Device: prototype of sensor
- ventilator (Active Comparator): The patient is his own control
  Interventions: Device: prototype of sensor

INTERVENTIONS:
Device: prototype of sensor — The investigational device is composed of a sensor placed on the respiratory line of the ventilated patients and connected to a ventilation measure unit which records the ventilation parameters

SUMMARY:
Recently, the threat of viral pandemics (Covid-19, severe acute respiratory syndrome, avian flu H5N1, and H1N1), which might result in thousands of patients requiring mechanical ventilation, has accelerated the need for mechanical ventilation equipment. Disaster may create thousands of critically ill patients requiring mechanical ventilation and may force difficult allocation decisions when demand greatly exceeds supply. Creating a new monitor will only add one more product to the one already used and create confusion for the user. Therefore, the aim is now to develop an independent ventilation module, compatible with the already existing cardiac monitors, which integrates advanced ventilation monitoring functions (mechanical ventilation and RCP). This module could be used by the teams already equipped with multiparametric monitors and be a real added value as the monitoring of the ventilation is critical, especially in emergency situations. Then, it could answer to the clinical need and massively equip every hospital care center in the event of mass casualty incident or viral pandemic. Moreover, this device could be used by emergency teams during daily operations. The aim of this study is to validate a prototype of sensor intended to monitor ventilator parameters of ventilated patients and guide healthcare professionals to provide safe ventilation.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patient aged 18 years or above
2. Patient ventilated with the reference ventilators: Servo U - Maquet Critical Care AB, Röntgenvägen 2, 171 54 Solna, Sweden for intensive care unit or Perseus - Drägerwerk AG & Co. KGaA, Moislinger Allee 53-55, 23542 Lübeck, Germany for operating room
3. Sedated patient with or without NBA (Neuromuscular Blocking Agent)
4. Patient with a positive end-expiratory pressure (PEEP) ≤ 10 cm H2O
5. Patient stable without recent (less than one hour) or planned intervention (such a bronchoscopy, prone positioning, physiotherapy)
6. The primary attending physician approves use of the protocol on the patient
7. Anticipated length of intubation > 2 hours per patient
8. The patient or legally authorized representative has signed and dated a written Informed Consent Form (ICF) prior to the initiation of any clinical investigation procedures
9. Patient affiliated to the French social security regimen
10. Procedure will be performed at least 30 minutes after inhaled treatment (eg salbutamol)

Exclusion Criteria:

1. Patient with a serious disease, for which the ventilation unplugging during a few seconds could have a serious impact (particularly patients with PaO2/Fi02 < 150 with pH < 7,30, with PEEP > 10 cm H20, or with Fi02 > 50%)
2. Patient with disease judged by the investigator to be incompatible with the conduct of the clinical investigation procedures or the interpretation of the clinical investigation results (example: IG-bronchopleural fistula)
3. Patient with a significant lower airway obstruction (asthma…), confirmed by ventilator spirometry.
4. Inability to maintain the airway intubation
5. Patient with a recent history of cardiac and/or respiratory arrest
6. Patient with multiple-organ system failure
7. Patient with hemodynamic instability (tachycardia, rapid change of vasopressor)
8. Pregnancy
9. Participation in another clinical investigation at the same time as the present clinical investigation
10. Nitric oxide use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2023-09-26 (Actual); Primary Completion 2024-06-06 (Actual); Study Completion 2024-06-06 (Actual)

PRIMARY OUTCOMES:
Number and proportion of patients for whom the insufflated volume measured by the sensor prototype is equivalent to the one measured by the ventilatory monito | 2 hours

SECONDARY OUTCOMES:
Number and proportion of patients for whom the exhaled volume measured by the sensor prototype are equivalent to the one measured by the ventilatory monitor | 2 hours
Number and proportion of patients for whom the pressure measured by the sensor prototype are equivalent to the one measured by the ventilatory monitor | 2 hours
Number and proportion of patients for whom the flow rate measured by the sensor prototype are equivalent to the one measured by the ventilatory monitor | 2 hours
Precision range of the insufflated volume between the sensor prototype and the one measured by the reference ventilator | 2 hours
Number and proportion of patients for whom the leak percentage calculated by the sensor prototype are equivalent to the one calculated by the ventilatory monitor ventilator | 2 hours
Number and proportion of patients for whom the insiratory time calculated by the sensor prototype are equivalent to the one calculated by the ventilatory monitor ventilator | 2 hours
Number and proportion of patients for whom the expiratory time calculated by the sensor prototype are equivalent to the one calculated by the ventilatory monitor ventilator | 2 hours
Number and proportion of patients for whom the pause time calculated by the sensor prototype are equivalent to the one calculated by the ventilatory monitor ventilator | 2 hours
Number and proportion of patients for whom the plateau time calculated by the sensor prototype are equivalent to the one calculated by the ventilatory monitor ventilator | 2 hours
Number and proportion of patients for whom the respiratory rate calculated by the sensor prototype are equivalent to the one calculated by the ventilatory monitor ventilator | 2 hours
Number and proportion of patients for whom the mechanical power calculated by the sensor prototype are equivalent to the one calculated by the ventilatory monitor ventilator | 2 hours
Number and proportion of patients for whom the lung resistance calculated by the sensor prototype are equivalent to the one calculated by the ventilatory monitor ventilator | 2 hours
Number and proportion of patients for whom the lung compliance calculated by the sensor prototype are equivalent to the one calculated by the ventilatory monitor ventilator | 2 hours
Number and proportion of patients for whom the lung elastance calculated by the sensor prototype are equivalent to the one calculated by the ventilatory monitor ventilator | 2 hours
Number and frequency of device deficiencies | 2 hours 30 minutes
Number and frequency of adverse events | 2 hours 30 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Besançon, Besançon, France

IPD SHARING:
Plan to Share IPD: No